CLINICAL TRIAL: NCT02921295
Title: A Comparative Analysis Between College Park Sidekick Feet and Conventional Stubby Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angela DeCandia (Other)
Collaborators: College Park Industries (Unknown)
Responsible Party: Sponsor-Investigator, Angela DeCandia, Prosthetic & Orthotic Resident, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO16050355
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-04

CONDITIONS: Amputation Stumps

ARMS (1):
- Sidekick Stubbies (Active Comparator): Conventional Stubby prostheses were used for baseline measures. In the sequential crossover design, articulated stubby prostheses ("Sidekick" manufactured by College Park Ind.) were used as intervention
  Interventions: Device: Sidekick Stubbies

INTERVENTIONS:
Device: Sidekick Stubbies

SUMMARY:
The purpose of this study is to compare the College Park Sidekicks to conventional stubby prosthetics to investigate their effects on bilateral above-knee-amputee gait velocity, exertion, and balance. The investigators aim to demonstrate that: (i) greater balance will be observed and reported on a level and gravel surface with the Sidekicks; (ii) time to complete the 10-meter walk test will be decreased wearing Sidekicks compared to the conventional stubby prosthesis; and (iii) subjects will report feeling less exerted with the sidekicks.

ELIGIBILITY:
Inclusion Criteria:

* bilateral transfemoral amputee
* own a pair of conventional stubby prosthesis with standard adaptation

Exclusion Criteria:

* dependence on assistive walking device or wheelchair (may use devices occasionally but should be able to ambulate without them)
* use of prosthesis that do not allow change of feet with standard adapters
* any medical condition that may put an individual in greater risk of injury than normal daily activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bakery Square MSPO labs, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequential Change of Intervention: Conventional Stubby prostheses and Sidekicks prostheses were used in a randomized sequence
Period: Sidekicks
Arm/Group | Sequential Change of Intervention
Started | 1
Completed | 1
Not Completed | 0
Period: Conventional Prostheses
Arm/Group | Sequential Change of Intervention
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequential Change of Interventions: Conventional Stubby prostheses will be used in this intervention
Arm/Group | Sequential Change of Interventions
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Speed for 10 Meter Walk Test
Description: The participant is timed while covering a 10-m distance unassisted (running start). The average speed is then calculated for each pass (one with each set of prosthetic feet), using the equation 10m/(recorded time in seconds). The average speed is computed as it is more reliable and representative than the instantaneous gait speed that may not be consistently maintained during the 10-m walk.
Time Frame: 2 times throughout study completion (every 1 hour during the 2 hour protocol)
Measure: Number; unit: m/s
Groups:
- Stubbies: Conventional Stubby prostheses as control intervention in cross-over trial
- Sidekicks: Active intervention in cross-over trial
Arm/Group | Stubbies | Sidekicks
Number analyzed (Participants) | 1 | 1
m/s | 0.57 | 0.53

2. Secondary Outcome: Timed up and go Test Time
Description: The test, as described in the protocol form, is performed three times with each intervention. This allows averaging to reduce the risk of random errors in timing the exercise. Accordingly, the participant is asked to repeat (with resting breaks in between) the tests three times with the stubbies and three times with the sidekicks.
Time Frame: 6 times throughout study completion (3 every 1 hour during the 2 hour protocol)
Measure: Mean (Standard Deviation); unit: s
Groups:
- Stubbies: control intervention
- Sidekicks: active intervention
Arm/Group | Stubbies | Sidekicks
Number analyzed (Participants) | 1 | 1
s | 0.27 (0.0103) | 0.25 (0.0074)

3. Secondary Outcome: Gait Symmetry Index
Description: Left/Right Step Duration Ratio. Perfect gait symmetry would result in a ratio of 1.000. Any deviation would indicate that step lengths differ between legs, indicating a more or less pronounced limping. The measure is computed from the intermediary step sample of gait with each intervention. This allows averaging to reduce the risk of random errors in assessment. Step samples were extracted from walking trial data with the stubbies and with the sidekicks. Each walking trial contains more than 30 individual steps for analysis.
Time Frame: 2 times throughout study completion (every 1 hour during the 2 hour protocol)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stubbies | Sidekicks
Number analyzed (Participants) | 1 | 1
ratio | 1.046 (0.119) | 0.965 (0.113)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Stubbies | Sidekicks
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02921295/SAP_000.pdf
  • Informed Consent Form (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02921295/ICF_001.pdf
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02921295/Prot_003.pdf